CLINICAL TRIAL: NCT05258136
Title: Clinical Study on the Efficacy and Safety of Low-dose CD20 Monoclonal Antibody Injection in Preemptive Treatment of Lymphoproliferative Diseases After Allogeneic Hematopoietic Stem Cell Transplantation in Patients With EBV-HLH/CAEBV
Brief Title: Low-dose CD20 Monoclonal Antibody Injection in Preemptive Treatment of PTLD in Patients With EBV-HLH/CAEBV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBV reactivation
Record Dates: First submitted 2022-02-24; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: PTLD; CAEBV; HLH
Keywords: preemptive therapy, CD20 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV-DNA positive patients (Experimental): EBV-DNA positive patients
  Interventions: Drug: low-dose CD20 monoclonal antibody injection

INTERVENTIONS:
Drug: low-dose CD20 monoclonal antibody injection — To comprehend the efficacy and safety of low-dose CD20 monoclonal antibody injection in preemptive treatment of EBV positive lymphoproliferative diseases after allo-HSCT in patients with EBV-HLH and CAEBV

SUMMARY:
This is a clinical study on the efficacy and safety of low-dose CD20 monoclonal antibody injection in preemptive treatment of EBV positive lymphoproliferative diseases after allo-HSCT in patients with EBV-HLH and CAEBV

DETAILED DESCRIPTION:
Purpose: To comprehend the efficacy and safety of low-dose CD20 monoclonal antibody injection in preemptive treatment of EBV positive lymphoproliferative diseases after allo-HSCT in patients with EBV-HLH and CAEBV Study subjects: PTLD patients undergoing allo-HSCT with CAEBV or EBV-HLH met the following conditions: (1) EBV-DNA (PBMC or plasma) > 1000 copies/ml in peripheral blood after transplantation; (2) no PTLD symptoms; (3) presence of aGVHD or clinicians believe that RI treatment is not suitable, or EBV-DNA persists > 1000 copies/ml after RI; (4) EBV infected lymphocytes; (4) B cell infection, or B cell copy number higher than other cell lines by 2 logs.

Therapeutic regimen: CD20 monoclonal antibody injection 100 mg/m2 was intravenously infused once a week. It can be discontinued after EBV-DNA negative for 2 consecutive times. Total dose≤ 4 applications per patient

ELIGIBILITY:
Inclusion Criteria:

* PTLD patients undergoing allo-HSCT with CAEBV or EBV-HLH met the following conditions: (1) EBV-DNA (PBMC or plasma) > 1000 copies/ml in peripheral blood after transplantation; (2) no PTLD symptoms; (3) presence of aGVHD or clinicians believe that RI treatment is not suitable, or EBV-DNA persists > 1000 copies/ml after RI; (4) EBV infected lymphocytes; (4) B cell infection, or B cell copy number higher than other cell lines by 2 logs.

Exclusion Criteria:

* Patients with active infection except for EBV; Active hepatitis B or C (positive HBV-DNA or HCV-RNA) ; Known life-threatening allergic reactions to CD20 Monoclonal Antibody Injection or its preparation ingredients; Participate in other clinical studies.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA | 4 weeks
  Incidence of negative ebv-dna conversion
PTLD | 1 year
  Incidence of PTLD

CONTACTS AND LOCATIONS:
Overall Officials: Yan Cui, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China